CLINICAL TRIAL: NCT00269282
Title: Motivating Asthma Adherence in Urban Teens
Brief Title: Increasing Adherence to Asthma Medication in Urban Teens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Cynthia Rand, Ph.D., Professor of Medicine and Psychiatry/Director, The Johns Hopkins Adherence Research Center, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 321; R01HL079301 (NIH)
Record Dates: First submitted 2005-12-21; First posted 2005-12-23 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Self-Management (SM) (Standard Care Group)
  Interventions: Behavioral: Self-Management Training
- 2 (Experimental): Motivational Interviewing plus Self-Management Training (MI+SM)
  Interventions: Behavioral: Self-Management Training; Behavioral: Motivational Interviewing (MI)

INTERVENTIONS:
Behavioral: Self-Management Training — Asthma education and self-monitoring strategies
Behavioral: Motivational Interviewing (MI) — Motivational Interviewing (MI) is a promising interventional approach that uses a client-centered, non-directive approach for enhancing motivation to change health behaviors.
  Arms: 2

SUMMARY:
The purpose of this study is to determine the effectiveness of two home-based asthma interventions in increasing adherence to daily asthma controller medication.

DETAILED DESCRIPTION:
BACKGROUND:

Low-income, minority teenagers have disproportionately high rates of asthma morbidity, including excess risk of emergency department (ED) care, hospitalization, and death from asthma, compared to white adolescents. Research by this group and others has documented that non-adherence with asthma treatment regimens is common among high-risk, inner city families with asthma, and that this poor adherence with prescribed therapies plays a significant contributing role in asthma morbidity. Inner-city adolescents with asthma are at particular risk of non-adherence, yet this population remains understudied. While asthma self-management training has shown promise in achieving some improvement in adherence with asthma, there are few intervention studies explicitly targeting adolescents, particularly those in the inner-city. Urban children typically assume primary control over their asthma management during late childhood/early adolescence. At the same time, adolescents' efforts to achieve autonomy and peer-acceptance may result in increased health risk behaviors, including poor asthma self-management. Developmentally-appropriate asthma self-management interventions are needed that target the unique challenges of adolescence. Motivational Interviewing (MI) is a promising interventional approach that uses a client-centered, non-directive approach for enhancing motivation to change health behaviors. MI techniques are developmentally consistent with the needs of early adolescents. MI does not assume that health will be the most important factor motivating the teen, but rather acknowledges and incorporates other motivators that are within the context of the teen's life, thus this intervention strategy has the flexibility to adapt to the unique life circumstances and stressors faced by urban adolescents. We propose to evaluate the relative effectiveness of a MI-focused self-management intervention (MI+SM) compared to a self-management (SM) intervention containing asthma education and self-monitoring strategies in a sample of 226 children age 10-15 years treated for asthma in the ED. Our primary hypothesis is that the MI+SM, as compared to SM alone, will result in greater improvement in medication adherence at 3- and 6-months post-randomization, as measured by electronic medication monitoring. Secondary outcomes include self-reported medication adherence, symptoms free days, urgent health care utilization for asthma, and caregiver/adolescent quality of life.

DESIGN NARRATIVE:

Participants will be randomly assigned to 1) Self-Management (SM; Standard Care Group) or 2) Motivational Interviewing plus Self-Management Training (MI+SM; Intervention Group). The duration of the intervention condition will be 5 home visits over 2 months. Follow-up measures will be collected from families at 3- and 6-months post-randomization.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Baltimore City
* Diagnosis of asthma or reactive airway disease
* Current emergency department visit or hospitalization for asthma
* Prescribed a daily asthma controller medication

Exclusion Criteria:

* Plans to move outside of the Baltimore City area within 1 year from study entry
* Current participation in another asthma education study
* Families unwilling or unable to participate
* Families who were enrolled and participated in the pilot study

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 207 (Actual)
Dates: Start 2006-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Adherence to asthma controller therapy as measured by electronic medication monitoring | Measured at baseline, 3 months, and 6 months

SECONDARY OUTCOMES:
Number of symptom-free days | Measured at baseline, 3 months, and 6 months
Emergency department utilization and hospitalization | Measured at baseline, 3 months, and 6 months
Caregiver/adolescent quality of life | Measured at baseline, 3 months, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia S. Rand, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital Pediatric Emergency Department, Baltimore, Maryland, United States